CLINICAL TRIAL: NCT05945732
Title: A Prospective, Non-interventional Study (NIS) With Trastuzumab Deruxtecan For Patients With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer Accompanied By a Disease Registry of Patients Treated With Conventional Chemotherapy (DESTINY Breast Respond HER2-low Europe)
Brief Title: DESTINY Breast Respond HER2-low Europe
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DS8201-0005-NIS-MA
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Unresectable Breast Cancer; Metastatic Breast Cancer; HER2-low Expressing Breast Cancer
Keywords: Unresectable Breast Cancer; Metastatic Breast Cancer; HER2-low Expressing Breast Cancer; Trastuzumab Deruxtecan; Enhertu®
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Trastuzumab deruxtecan (T-DXd): Participants with HER2-low expressing unresectable and/or metastatic breast cancer who will be treated with trastuzumab deruxtecan and part of the enrolled participants will receive conventional chemotherapy. The participants on conventional chemotherapy will be analyzed exploratory only.
  Interventions: Drug: Trastuzumab deruxtecan

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — This is a non-interventional study and medication will be administered according to the SmPC as local standard of care and as part of the routine clinical practice.
  Trastuzumab (T-DXd) to be administered according to the SmPC.
  Conventional therapy (eg. capecitabine, eribulin, gemcitabine, paclitaxel, nab paclitaxel) to be administered according to the SmPC.
  Other Names: T-DXd

SUMMARY:
Trastuzumab deruxtecan (T-DXd) as monotherapy is indicated for the treatment of adult patients with unresectable or metastatic HER2-low breast cancer who have received prior chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.

DETAILED DESCRIPTION:
This non-interventional study will investigate the effectiveness withT-DXd, the demographic and clinical characteristics of the patients, treatment patterns, tolerability, management of adverse drug reactions (ADRs), and patient experience of T-DXd in patients with HER2-low unresectable and/or metastatic breast cancer. Patients will be treated according to the proposed indication statement in the Summary of Product Characteristics (SmPC). No drug product will be administered as part of this study.

Data on conventional chemotherapy (i.e., including but not limited to capecitabine, eribulin, gemcitabine, paclitaxel and nab-paclitaxel) will also be collected in a disease registry part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years) with histological or cytological confirmed diagnosis of unresectable and/or mBC
* Documented HER2-low status (IHC1+, IHC2+/ISH-)
* Patients who have received prior chemotherapy in the metastatic setting or patients who have developed disease recurrence during or within 6 months of completing adjuvant chemotherapy
* Decision to newly initiate therapy of T-DXd or conventional chemotherapy according to the physicians choice per SmPC
* Written and signed Informed Consent to participate in the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients who at time of data collection for this study are participating in or have participated in an interventional study that remains blinded.

No other specific exclusion criteria are defined, as patients will be treated according to the proposed indication statements in the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with unresectable or metastatic HER2-low breast cancer who have received prior chemotherapy in the metastatic setting or developed disease recurrence during or within 6 months of completing adjuvant chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1155 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Real World Time to Next Treatment (rwTTNT1) in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer | Baseline up to 31 months

SECONDARY OUTCOMES:
Type of Treatment Patterns in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer | Baseline up to 31 months
Number of Physician-reported Safety Events of Interest in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer (T-DXd only) | Baseline up to 31 months
Number of Participants Receiving Prophylactic and Reactive Treatment Management for Physician-reported Safety Events of Interest in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer (T-DXd only) | Baseline up to 31 months
Real World Time to Permanent Treatment Discontinuation (rwTTD1) in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer | Baseline up to 31 months
Patient's Global Impression of Treatment Tolerability (PGI-TT) in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer | Baseline up to 31 months
  The PGI-TT is designed to assess the treatment tolerability of the medicine. Participants will rate the bother associated with any treatment-related symptoms based on a 5-point scale ranging from 1 (not at all) to 5 (very much). Higher scores indicate a worse outcome.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Score in Participants With HER2-low Expressing Unresectable and/or Metastatic Breast Cancer | Baseline up to 31 months
  The EORTC QLQ-C30 questionnaire is designed to measure cancer patients' physical, psychological and social functions. The EORTC QLQ-C30 scales and single-item scales range in score from 0 to 100. A higher score for the functioning scales and global health status denotes a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Number of Participants Reporting Nausea and Vomiting as Assessed by a Patient Diary | Baseline up to 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company
Locations (210):
- Austria (14):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - LKH Hochsteiermark-Leoben, Leoben
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz
  - Interne II, LKH Feldkirch, Rankweil
  - KH der Barmherzigen Brüder Salzburg, Salzburg
  - Uniklinikum Salzburg, Salzburg
  - Medical University of Vienna, Vienna
  - Medizinische Universität Wien, Vienna
  - Krankenhaus Hietzing, Vienna
  - Salzkammergut Klinikum Vöcklabruck, Vöcklabruck
  - Klinikum Wels-Grieskirchen GmbH, Wels
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Belgium (16):
  - ASZ Aalst, Aalst
  - Chirec Delta Hospital, Auderghem
  - Imeldaziekenhuis Bonheiden, Bonheiden
  - AZ Klina, Brasschaat
  - AZ Sint-Jan Brugge av, Bruges
  - CHU Brugmann, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Chu Helora- Hôpital de La Louvière- site Jolimont, Haine-Saint-Paul
  - Jessa Ziekenhuis, Hasselt
  - CHU Tivoli, La Louvière
  - CHC MontLegia, Liège
  - Hôpital de la Citadelle, Liège
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
  - Clinique Saint Pierre Ottignies, Ottignies
  - VITAZ, Sint-Niklaas
  - CHR Verviers East Belgium, Verviers
- Denmark (6):
  - Aalborg Universitetshospital, Syd, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Herlev Hospital, Herlev
  - Onkologisk og Palliativ afdeling, Nordsjællands Hospital, Hillerød
  - Naestved Hospital, Næstved
  - Sygehus Sønderjylland, Sønderborg, Sønderborg
- France (66):
  - CHU Amiens Picardie, Amiens
  - Clinique de l'Europe, Amiens
  - Hôpital Privé d'Antony, Antony
  - Hôpital Privé les Bonnettes, Arras
  - Institut du Cancer Avignon Provence, Avignon
  - CH Cote Basque, Bayonne
  - Clinique Belharra, Bayonne
  - Chu Jean Minjoz Besancon, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - Centre hospitalier Fleyriat, Bourg-en-Bresse
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Metropole Savoie, Chambéry
  - Pole Sante Leonard De Vinci, Chambray-lès-Tours
  - CH Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Polyclinique St Côme, Compiègne
  - Hôpital Henri Mondor, Créteil
  - Centre Léonard de Vinci, Dechy
  - Centre Georges Francois Leclerc, Dijon
  - CHU Martinique, Fort de France Cedex
  - CHI Frejus Saint Raphael, Fréjus
  - Groupe Hospitalier Mutualiste (GHM) de Grenoble - Institut Daniel Hollard (IDH), Grenoble
  - Polyclinique De Blois, La Chaussée-Saint-Victor
  - La Tronche - CHU Grenoble, La Tronche
  - Centre de cancerologie de la Sarthe, Le Mans
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Hôpital Franco-Britannique Cognac Jay, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - CHU Lille, Lille
  - Hôpital Prive Le Bois, Lille
  - CHU de Limoges, Limoges
  - Hospices Civils De Lyon, Lyon
  - Hôpital Jean Mermoz, Lyon
  - Hôpital-Clinique Claude Bernard, Metz
  - GH Havre, Montivilliers
  - Clinique Clementville, Montpellier
  - Groupe Hospitalier privé Ambroise Pare Hartmann, Neuilly-sur-Seine
  - Hopital Americain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier de Niort, Niort
  - Centre Médical ONCOGARD, Nîmes
  - Institut Curie, Paris
  - Groupement Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hôpital Saint Joseph, Paris
  - Centre Hospitalier de Pau, Pau
  - CHU Poitiers, Poitiers
  - Institut Godinot, Reims
  - Polyclinique Courlancy, Reims
  - Centre Eugene Marquis, Rennes
  - Clinique Saint Hilaire, Rouen
  - Clinique Mathilde, Rouen
  - Saint Cloud -Rene Huguenin Institut Curie, Saint-Cloud
  - CHU Réunion Site Sud, Saint-Paul
  - Institut De Cancerologie Paris Nord, Sarcelles
  - Centre Hospitalier de Sens, Sens Cédex
  - Hôpital Foch, Suresnes
  - CHR Metz Thionville, Thionville
  - HIA Sainte-Anne, Toulon
  - Centre Hospitalier de Troyes, Troyes
  - Hopital Prive Drome Ardeche, Valence
  - Nouvelle Clinique Des Dentellières, Valenciennes
  - Institut De Cancerologie De Lorraine, Vandœuvre-lès-Nancy
  - Centre d'oncologie Saint-Yves, Vannes
  - Médipôle Hôpital Mutualiste, Villeurbanne
- Italy (33):
  - Azienda Ospedaliera di Alessandria, Alessandria
  - Ospedale SS Annunziata, Chieti
  - Ospedale Citta' di Castello USL Umbria 1, Città di Castello
  - Ospedale San Giuseppe - Azienda USL Toscana Centro, Empoli
  - ASL Lecce - Ospedale "Vito Fazzi", Lecce
  - ASST Lecco - PO "Alessandro Manzoni", Lecco
  - AULSS 9 Scaligera - Ospedale Mater Salutis, Legnago
  - ASST Ovest Milanese - Ospedale di Legnano, Legnano
  - Ospedale Generale Provinciale di Macerata, Macerata
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST IRCCS, Meldola
  - AOU di Modena, Modena
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - AOU Federico II, Napoli
  - AOU Maggiore della Carità di Novara, Novara
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua
  - La Maddalena S.p.A., Palermo
  - ARNAS Ospedale Civico e Benfratelli, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AOU Pisana - Stabilimento Santa Chiara, Pisa
  - AO Regionale San Carlo, Potenza
  - GOM "BMM" - Presidio Ospedaliero Morelli, Reggio Calabria
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - ASL RM 2 Ospedale Pertini, Roma
  - AO San Giovanni Addolorata, Roma
  - AOU "San Giovanni di Dio e Ruggi d'Aragona", Salerno
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - AOU Sassari - Ospedale Civile SS. Annunziata, Sassari
  - Ospedale San Vincenzo, Taormina
  - AOU Città della Salute e della Scienza di Torino - Ospedale Molinette, Torino
  - AO Ordine Mauriziano, Torino
  - AULSS n. 2 Marca trevigiana - Ospedale "Cà Foncello", Treviso
  - ASUFC Udine - Santa Maria della Misericordia, Udine
  - ASST Sette Laghi "Ospedale di Circolo e Fondazione Macchi ", Varese
- Norway (5):
  - Nordlandssjukhuset Bodø, Bodø
  - Drammen Sykehus, Drammen
  - Sørlandet sykehus / Kristiansand Hospital, Kristiansand
  - Sykehuset Telemark, Skien
  - Universitetssjukhuset Nord-Norge, Tromsø
- Portugal (12):
  - Hospital de Cascais, Alcabideche, Lisboa
  - ULS Amadora Sintra, Amadora, Lisboa
  - ULS Braga, Braga
  - IPO Lisboa, Lisbon
  - Dra. Berta Sousa, Lisbon
  - Hospital da Luz Lisboa, Lisbon
  - ULS Santa Maria, Lisbon
  - ULS Loures-Odivelas - Hospital Beatriz Ângelo, Loures
  - ULS Santo António, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, Porto
  - ULS Matosinhos, Porto
  - ULS Trás-os-Montes e Alto Douro, Vila Real
- Spain (37):
  - Hospital Clinico Universitario de Albacete, Albacete
  - Hospital Universitario de La Ribera, Alzira
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario de Puerto Real, Cadiz
  - Hospital Universitario San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario de Elche, Elche
  - Hospital de Galdakao, Galdakao
  - Hospital Clinico Universitario de Granada (PTS), Granada
  - Hospital Universitario Médico-Quirúrgico de Jaén, Jaén
  - Complejo Asistencial Universitario de León, León
  - Hospital Universitario San Pedro de Logroño, Logroño
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario la Princesa, Madrid
  - Hospital MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital de Getafe, Madrid
  - Hospital Virgen Arrixaca de Murcia, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Asistencial Universitario de Palencia, Palencia
  - Hospital Son Llatzer, Palma
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Pontevedra, Pontevedra
  - Hospital San Joan de Reus, Reus
  - Hospital Universitari Parc Taulí, Sabadell
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario General de Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitario Rio Hortega, Valladolid
  - Complejo Hospitalario Universitario De Vigo, Vigo Pontevedra
- Sweden (9):
  - Onkologikliniken Mälarsjukhuset, Eskilstuna
  - Gävle Hospital, Gävle
  - Ryhov County Hospital, Jönköping
  - Department of Oncology, Örebro University Hospital, Örebro
  - Capio St Görans sjukhus, Stockholm
  - Bröstcentrum, Karolinska Universitetssjukhuset Solna, Stockholm
  - Onkologkliniken Sundsvalls Sjukhus, Sundsvall
  - Cancercentrum, Norrlands Universitetssjukhus, Umeå
  - Department of Oncology, Västerås, Västerås
- Switzerland (12):
  - Kantonsspital Baden, Baden
  - Spital Thurgau AG - Kantonsspital Frauenfeld, Frauenfeld
  - Centre du sein Fribourg, Fribourg
  - Clinique Generale-Beaulieu / Clinique de Genolier, Geneva
  - Réseau Hospitalier Neuchâtelois (RHNe), La Chaux-de-Fonds
  - Réseau du Sein Lausanne, Lausanne
  - CHUV, Lausanne
  - Kantonsspital Baselland, Liestal
  - Kantonsspital St.Gallen, Sankt Gallen
  - Hôpital du Valais Sion, Sion
  - ZIO AG, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guarneri V, Passos Coelho JL, Duhoux FP, Egle D, Garcia-Saenz JA, Penault-Llorca F, Selander K, Wildiers H, Zaman K, Laeis P, Lucerna M, Pierga JY. Study design for DESTINY-Breast Respond HER2-low Europe: T-DXd in patients with HER2-low advanced breast cancer. Future Oncol. 2024;20(18):1237-1250. doi: 10.2217/fon-2024-0015. Epub 2024 Apr 9. PMID 38592002